CLINICAL TRIAL: NCT06917001
Title: A Randomized, Double-blind, Placebo-controled, Phase 2a Trial Evaluating the Safety and Initial Efficacy of Resomelagon in Patients With Dengue Infection
Brief Title: Clinical Trial Evaluating Safety and Efficacy of Resomelagon on Dengue Infection (RESOVIR-2)
Acronym: RESOVIR-2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Instituto Nacional de Ciência e Tecnologia em Dengue (INCT em Dengue) (Unknown)
Responsible Party: Principal Investigator, Mauro Martins Teixeira, Pricipal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 85788125.5.1001.5415
Record Dates: First submitted 2025-03-20; First posted 2025-04-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Dengue Fever
Keywords: Resomelagon; Resolution of inflammation; Melanocortin; Dengue; RESOVIR-2
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resomelagon (Experimental): Resomelagon, 100mg, orally, once daily plus standard treatment
  Interventions: Drug: Resomelagon; Other: Standard Treatment
- Placebo (Placebo Comparator): Placebo plus standard treatment
  Interventions: Drug: Placebo; Other: Standard Treatment

INTERVENTIONS:
Drug: Resomelagon — Resomelagon 100mg, orally, once daily.
  Arms: Resomelagon
Drug: Placebo — Placebo
  Arms: Placebo
Other: Standard Treatment — Hydration and symptomatic therapy as indicated for Dengue fever.

SUMMARY:
The goal of this clinical trial is to understand if Resomelagon can treat adult patients with Dengue virus infection. The main questions the investigators aim to answer are:

Is Resomelagon safe to use in patients with Dengue? Is Resomelagon able to reduce the duration of illness? (defined by clinical and laboratory criteria) Participants will be allocated to Resomelagon or placebo groups in this study and asked to take the medication and submitted to blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 to 65 years old;
* Able to understand study procedures and give informed consent;
* Presents with more than 36 and less than 84h since symptoms onset;
* Symptoms compatible with dengue infection (fever, myalgia, arthralgia, headache or conjunctivitis) with positive antigen test or polymerase chain reaction test.

Exclusion Criteria:

* Has any comorbidity which is perceived as significant by the investigator;
* Significant laboratory abnormalities discovered at triage: Hemoglobin <10g/dL; Platelet count < 50.000/microL; alanine transaminase > 3x upper limit of normal; Total bilirubin >1,5 x upper limit of normal; glomerular filtration rate < 60mls/min/1,73m2;
* Contraindications or known hypersensitivity to Resomelagon;
* Presents as dengue with warning signs or severe dengue at inclusion;
* Currently participating in another drug clinical trial;
* Clinical evidence of another infection that might explain current symptoms;
* Pregnant women or women actively trying to achieve pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety of Resomelagon in Dengue patients | 28 days
  Incidence of clinical or laboratory adverse events. All symptoms, illness and laboratory abnormalities will be graded by the investigators in accordance to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse events graded 3 or more in severity will be registered. Serious adverse events will be reported and registered. Incidence of adverse events will be compared between placebo and intervention groups.
Efficacy of Resomelagon in decreasing illness duration | 10 days
  Time to resolution of illness as defined by a composite outcome:
  Patient afebrile for 48 hours without paracetamol (or other drugs to treat fever) ingestion; Rising platelet counts of >20% of the lowest, or normal platelet counts if the patient did not have thrombocytopenia, following two consecutive measurements from the lowest platelet count Haematocrit stabilized or return to the normal hematocrit for age & sex, following two consecutive measurements Absence of bleeding or significant vomiting for 48h.

SECONDARY OUTCOMES:
Efficacy of Resomelagon in reducing illness Severity | 10 days
  Incidence of dengue with warning signs or severe dengue in the study patients
Efficacy of Resomelagon in reducing plasma leakage | 10 days
  Incidence of hemoconcentration (hematocrit increase of >10% from inclusion or elevated for age & sex) OR evidence of pleural effusion OR evidence of ascitis OR pericardial effusion
Efficacy of Resomelagon in reducing dengue hospitalization or prolonged observation in the Emergency department | 10 days
  Incidence of a stay of more than 12h in the emergency department or hospital admission

OTHER OUTCOMES:
Evaluation of proinflammatory cytokines. | 28 days
  Measurement of proinflammatory cytokines using Meso Scale Discovery (MSD) platform with V-Plex proinflammatory panel 1 (Human).
Evaluation of proinflammatory chemokines. | 28 days
  Measurement of proinflammatory chemokines using Meso Scale Discovery (MSD) platform with V-Plex Chemokine Panel 1 (Human).
Evaluation of cytokine production by mononuclear cells. | 28 days
  Mononuclear cells from peripheral blood will be evaluated by flow cytometry for assessment of their surface inflammatory biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro M Teixeira, MD PhD, Principal Investigator — Federal University of Minas Gerais
Locations (2):
- Brazil (2):
  - Clinical Research Unit, Belo Horizonte, Minas Gerais
  - Centro Integrado de Pesquisa, São José do Rio Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Almeida PRJ, Periard AM, Tana FL, Avila RE, Milhorato LB, Alcantara KMM, Resende CB, Serufo AV, Santos FR, Teixeira DC, Queiroz-Junior CM, Fonseca TCM, Silva BLV, Costa VV, Souza RP, Perretti M, Jonassen TEN, Teixeira MM. Effects of a pro-resolving drug in COVID-19: preclinical studies to a randomized, placebo-controlled, phase Ib/IIa trial in hospitalized patients. Br J Pharmacol. 2024 Dec;181(23):4750-4765. doi: 10.1111/bph.17322. Epub 2024 Aug 19. PMID 39159951
- [Result] Ehteshami M, Tao S, Zandi K, Hsiao HM, Jiang Y, Hammond E, Amblard F, Russell OO, Merits A, Schinazi RF. Characterization of beta-d-N4-Hydroxycytidine as a Novel Inhibitor of Chikungunya Virus. Antimicrob Agents Chemother. 2017 Mar 24;61(4):e02395-16. doi: 10.1128/AAC.02395-16. Print 2017 Apr. PMID 28137799
- [Result] An YJ, Choi SM, Choi ER, Nam YE, Seo EW, Ahn SB, Jang Y, Kim M, Cho JH. Synthesis and biological evaluation of new beta-D-N4-hydroxycytidine analogs against SARS-CoV-2, influenza viruses and DENV-2. Bioorg Med Chem Lett. 2023 Mar 1;83:129174. doi: 10.1016/j.bmcl.2023.129174. Epub 2023 Feb 8. PMID 36764470
- [Result] Imran M, Kumar Arora M, Asdaq SMB, Khan SA, Alaqel SI, Alshammari MK, Alshehri MM, Alshrari AS, Mateq Ali A, Al-Shammeri AM, Alhazmi BD, Harshan AA, Alam MT, Abida. Discovery, Development, and Patent Trends on Molnupiravir: A Prospective Oral Treatment for COVID-19. Molecules. 2021 Sep 24;26(19):5795. doi: 10.3390/molecules26195795. PMID 34641339
- [Result] Singh AK, Singh A, Singh R, Misra A. Molnupiravir in COVID-19: A systematic review of literature. Diabetes Metab Syndr. 2021 Nov-Dec;15(6):102329. doi: 10.1016/j.dsx.2021.102329. Epub 2021 Oct 30. PMID 34742052
- [Result] Silva MMO, Kikuti M, Anjos RO, Portilho MM, Santos VC, Goncalves TSF, Tauro LB, Moreira PSS, Jacob-Nascimento LC, Santana PM, Campos GS, Siqueira AM, Kitron U, Reis MG, Ribeiro GS. Risk of chronic arthralgia and impact of pain on daily activities in a cohort of patients with chikungunya virus infection from Brazil. Int J Infect Dis. 2021 Apr;105:608-616. doi: 10.1016/j.ijid.2021.03.003. Epub 2021 Mar 5. PMID 33684559
- [Result] Dengue Alliance. Electronic address: gnmalavige@dndi.org; Dengue Alliance. Treatments for dengue: a Global Dengue Alliance to address unmet needs. Lancet Glob Health. 2023 Nov;11(11):e1680-e1681. doi: 10.1016/S2214-109X(23)00362-5. Epub 2023 Aug 31. No abstract available. PMID 37660714
- [Result] Utarini A, Indriani C, Ahmad RA, Tantowijoyo W, Arguni E, Ansari MR, Supriyati E, Wardana DS, Meitika Y, Ernesia I, Nurhayati I, Prabowo E, Andari B, Green BR, Hodgson L, Cutcher Z, Rances E, Ryan PA, O'Neill SL, Dufault SM, Tanamas SK, Jewell NP, Anders KL, Simmons CP; AWED Study Group. Efficacy of Wolbachia-Infected Mosquito Deployments for the Control of Dengue. N Engl J Med. 2021 Jun 10;384(23):2177-2186. doi: 10.1056/NEJMoa2030243. PMID 34107180
- [Result] Schilling WHK, Jittamala P, Watson JA, Boyd S, Luvira V, Siripoon T, Ngamprasertchai T, Batty EM, Cruz C, Callery JJ, Singh S, Saroj M, Kruabkontho V, Ngernseng T, Tanglakmankhong N, Tubprasert J, Abdad MY, Madmanee W, Kouhathong J, Suwannasin K, Pagornrat W, Piaraksa N, Hanboonkunupakarn P, Hanboonkunupakarn B, Poovorawan K, Potaporn M, Srisubat A, Loharjun B, Taylor WRJ, Chotivanich V, Chotivanich K, Imwong M, Pukrittayakamee S, Dondorp AM, Day NPJ, Teixeira MM, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Antiviral efficacy of molnupiravir versus ritonavir-boosted nirmatrelvir in patients with early symptomatic COVID-19 (PLATCOV): an open-label, phase 2, randomised, controlled, adaptive trial. Lancet Infect Dis. 2024 Jan;24(1):36-45. doi: 10.1016/S1473-3099(23)00493-0. Epub 2023 Sep 28. PMID 37778363
- [Result] Jittamala P, Schilling WHK, Watson JA, Luvira V, Siripoon T, Ngamprasertchai T, Almeida PJ, Ekkapongpisit M, Cruz C, Callery JJ, Boyd S, Anunsittichai O, Hongsuwan M, Singhaboot Y, Pagornrat W, Tuntipaiboontana R, Kruabkontho V, Ngernseng T, Tubprasert J, Abdad MY, Keayarsa S, Madmanee W, Aguiar RS, Santos FM, Batty EM, Hanboonkunupakarn P, Hanboonkunupakarn B, Sookprome S, Poovorawan K, Imwong M, Taylor WRJ, Chotivanich V, Sangketchon C, Ruksakul W, Chotivanich K, Pukrittayakamee S, Dondorp AM, Day NPJ, Teixeira MM, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Clinical Antiviral Efficacy of Remdesivir in Coronavirus Disease 2019: An Open-Label, Randomized Controlled Adaptive Platform Trial (PLATCOV). J Infect Dis. 2023 Nov 11;228(10):1318-1325. doi: 10.1093/infdis/jiad275. PMID 37470445
- [Result] Butler CC, Hobbs FDR, Gbinigie OA, Rahman NM, Hayward G, Richards DB, Dorward J, Lowe DM, Standing JF, Breuer J, Khoo S, Petrou S, Hood K, Nguyen-Van-Tam JS, Patel MG, Saville BR, Marion J, Ogburn E, Allen J, Rutter H, Francis N, Thomas NPB, Evans P, Dobson M, Madden TA, Holmes J, Harris V, Png ME, Lown M, van Hecke O, Detry MA, Saunders CT, Fitzgerald M, Berry NS, Mwandigha L, Galal U, Mort S, Jani BD, Hart ND, Ahmed H, Butler D, McKenna M, Chalk J, Lavallee L, Hadley E, Cureton L, Benysek M, Andersson M, Coates M, Barrett S, Bateman C, Davies JC, Raymundo-Wood I, Ustianowski A, Carson-Stevens A, Yu LM, Little P; PANORAMIC Trial Collaborative Group. Molnupiravir plus usual care versus usual care alone as early treatment for adults with COVID-19 at increased risk of adverse outcomes (PANORAMIC): an open-label, platform-adaptive randomised controlled trial. Lancet. 2023 Jan 28;401(10373):281-293. doi: 10.1016/S0140-6736(22)02597-1. Epub 2022 Dec 22. PMID 36566761
- [Result] Schilling WHK, Jittamala P, Watson JA, Ekkapongpisit M, Siripoon T, Ngamprasertchai T, Luvira V, Pongwilai S, Cruz C, Callery JJ, Boyd S, Kruabkontho V, Ngernseng T, Tubprasert J, Abdad MY, Piaraksa N, Suwannasin K, Hanboonkunupakarn P, Hanboonkunupakarn B, Sookprome S, Poovorawan K, Thaipadungpanit J, Blacksell S, Imwong M, Tarning J, Taylor WRJ, Chotivanich V, Sangketchon C, Ruksakul W, Chotivanich K, Teixeira MM, Pukrittayakamee S, Dondorp AM, Day NPJ, Piyaphanee W, Phumratanaprapin W, White NJ; PLATCOV Collaborative Group. Pharmacometrics of high-dose ivermectin in early COVID-19 from an open label, randomized, controlled adaptive platform trial (PLATCOV). Elife. 2023 Feb 21;12:e83201. doi: 10.7554/eLife.83201. PMID 36803992
- [Result] Hammond J, Leister-Tebbe H, Gardner A, Abreu P, Bao W, Wisemandle W, Baniecki M, Hendrick VM, Damle B, Simon-Campos A, Pypstra R, Rusnak JM; EPIC-HR Investigators. Oral Nirmatrelvir for High-Risk, Nonhospitalized Adults with Covid-19. N Engl J Med. 2022 Apr 14;386(15):1397-1408. doi: 10.1056/NEJMoa2118542. Epub 2022 Feb 16. PMID 35172054
- [Result] Chen P, Nirula A, Heller B, Gottlieb RL, Boscia J, Morris J, Huhn G, Cardona J, Mocherla B, Stosor V, Shawa I, Adams AC, Van Naarden J, Custer KL, Shen L, Durante M, Oakley G, Schade AE, Sabo J, Patel DR, Klekotka P, Skovronsky DM; BLAZE-1 Investigators. SARS-CoV-2 Neutralizing Antibody LY-CoV555 in Outpatients with Covid-19. N Engl J Med. 2021 Jan 21;384(3):229-237. doi: 10.1056/NEJMoa2029849. Epub 2020 Oct 28. PMID 33113295
- [Result] Weinreich DM, Sivapalasingam S, Norton T, Ali S, Gao H, Bhore R, Musser BJ, Soo Y, Rofail D, Im J, Perry C, Pan C, Hosain R, Mahmood A, Davis JD, Turner KC, Hooper AT, Hamilton JD, Baum A, Kyratsous CA, Kim Y, Cook A, Kampman W, Kohli A, Sachdeva Y, Graber X, Kowal B, DiCioccio T, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD; Trial Investigators. REGN-COV2, a Neutralizing Antibody Cocktail, in Outpatients with Covid-19. N Engl J Med. 2021 Jan 21;384(3):238-251. doi: 10.1056/NEJMoa2035002. Epub 2020 Dec 17. PMID 33332778
- [Result] Gottlieb RL, Vaca CE, Paredes R, Mera J, Webb BJ, Perez G, Oguchi G, Ryan P, Nielsen BU, Brown M, Hidalgo A, Sachdeva Y, Mittal S, Osiyemi O, Skarbinski J, Juneja K, Hyland RH, Osinusi A, Chen S, Camus G, Abdelghany M, Davies S, Behenna-Renton N, Duff F, Marty FM, Katz MJ, Ginde AA, Brown SM, Schiffer JT, Hill JA; GS-US-540-9012 (PINETREE) Investigators. Early Remdesivir to Prevent Progression to Severe Covid-19 in Outpatients. N Engl J Med. 2022 Jan 27;386(4):305-315. doi: 10.1056/NEJMoa2116846. Epub 2021 Dec 22. PMID 34937145

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT06917001/Prot_SAP_000.pdf